CLINICAL TRIAL: NCT00313235
Title: Combined Modality Treatment for Patients With Stage IV Melanoma: Cyclophosphamide and a Dendritic Cell Vaccine Loaded With Killed Allogeneic Melanoma Cells
Brief Title: Combined Modality Treatment for Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Baylor IRB #006-025-01; IND 12919 (Other: FDA-CBER)
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Malignant Melanoma Stage IV
Keywords: Dendritic Vaccine; Melanoma; Cyclophosphamide (CPA)
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DC Vaccine and Cyclophosphamide (Experimental): Autologous dendritic cells (DC) are derived from PBMC, cultured with cytokines, pulsed ex vivo with irradiated allogeneic (Colo 829) melanoma cells. About 15 x 10^6 dendritic cells will be injected subcutaneously, in 3 separate sites (3.3 ml/site).
  Patients will receive a total of 7 doses of the vaccination. Each individual dose will be administered at weeks: 0, 2, 4, 6, 11, 14, and 18. Patients with SD, PR according to RECIST criteria may receive 4 more vaccines at 36, 48, 60 and 72 weeks. Patients with CR will receive 4 additional vaccines at 36, 48, 72, and 96 weeks.
  CPA will be administered 300mg/m2, intravenously over a 2-hour infusion 24 hours prior to DC vaccinations # 1, 3, 5, 6 and 7. Frequency of CPA administration might be increased based on their T cell measure.
  Interventions: Biological: DC Vaccine and Cyclophosphamide

INTERVENTIONS:
Biological: DC Vaccine and Cyclophosphamide — Autologous dendritic cells (DC) are derived from PBMC, cultured with cytokines, pulsed ex vivo with irradiated allogeneic (Colo 829) melanoma cells. About 15 x 10^6 dendritic cells will be injected subcutaneously, in 3 separate sites (3.3 ml/site).
  Patients will receive a total of 7 doses of the vaccination. Each individual dose will be administered at weeks: 0, 2, 4, 6, 11, 14, and 18. Patients with SD, PR according to RECIST criteria may receive 4 more vaccines at 36, 48, 60 and 72 weeks. Patients with CR will receive 4 additional vaccines at 36, 48, 72, and 96 weeks.
  CPA will be administered 300mg/m2, intravenously over a 2-hour infusion 24 hours prior to DC vaccinations # 1, 3, 5, 6 and 7. Frequency of CPA administration might be increased based on their T cell measure.
  Other Names: Cyclophosphamide - CPA; Dendritic Cell Vaccine - DC Vaccine

SUMMARY:
The purpose of this study is to test a combined treatment using cyclophosphamide and a novel dendritic cell vaccine in patients with Stage IV melanoma.

DETAILED DESCRIPTION:
A novel dendritic cell vaccine is being developed at the Baylor Institute for Immunology Research. Pre-clinical studies have found that this dendritic cell vaccine is more efficient in inducing a tumor specific immunity than other dendritic cell vaccines. Further studies in BIIR have been done with dendritic cells that were loaded with killed melanoma cells from a melanoma cell line treated with heat before loading. Both studies have shown that DCs manufactured in this novel way were more efficient in priming the melanoma specific CD8+ cells. Our previous studies indicate that a portion of patients with stage IV melanoma cannot mount an immune response to tumor antigens presented on dendritic cells. Also, regulatory/suppressor T cells can be identified in the blood of these patients, which may account for the lack of induction of T cell immunity to dendritic cell vaccines. Cyclophosphamide treatments have improved antitumor immunity in humans with melanoma and a clear relationship between cyclophosphamide dosage and suppressor cell activity has been documented. Therefore, this trial will test a combined modality treatment, using dendritic cell based vaccines in patients who have been treated with cyclophosphamide.

This clinical trial will evaluate the cyclophosphamide/dendritic cell vaccine in patients with Stage IV melanoma. The trial will accrue a total of 33 subjects. The primary goal of this trial will be to test the safety/tolerability/feasibility of the combined modality and the rate of objective clinical response.However if feasibility data in the first 10 subjects demonstrate the need to adjust the dose of CPA, the new dose will be tested in the next 10 subjects thereby extending the accrual to 43 subjects. A 15% objective response rate will be accepted in patients with stage IV Melanoma.

Patients will receive cyclophosphamide 300 mg/m2, administered 24 hours prior to DC vaccinations # 1, 3, 5, 6 and 7. Each subject will initially receive 7 doses of vaccination with each individual dose being administered at weeks 0, 2, 4, 6, 10, 14 and 18. A clinical evaluation of the patients will be done at weeks 10 & 20. Patients with progressive disease will be taken off of the study. Patients with SD, PR or CD (according to RECIST criteria) may receive 4 more vaccinations. Scans and re-staging tests will be performed at scheduled intervals throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Stage M1a, M1b, M1c biopsy proven metastatic melanoma.
* Ages 21-75.
* Karnofsky performance status greater than/equal to 80%.
* Measurable metastatic lesions by physical exam or scans.
* Acceptable CBC and blood chemistry results.
* Adequate hepatic and renal function.
* No active CNS metastatic disease. If CNS history is present, lesions must have been resected by surgery and/or gamma knife irradiation at least 3 months prior to study entry. The total number of CNS lesions at diagnosis should not exceed 3.
* Written informed consent.

Exclusion Criteria:

* Patients that have received more than 8 cycles of chemotherapy for metastatic melanoma.
* Patients who have received chemotherapy less than 4 weeks before beginning the trial.
* Patients who have received IFN alpha-2b or GM-CSF less than 4 weeks before beginning the trial.
* Patients who have received high-dose IL-2 less than 4 weeks before beginning the trial.
* Patients diagnosed with more than 3 CNS metastatic melanoma lesions.
* More than 5 hepatic lesions or any hepatic lesion larger than 5 cm.
* Baseline serum LDH greater than 1.1 times the upper limit of normal.
* Patients who are HIV positive.
* Patients who are pregnant.
* Patients who have receive corticosteroids or other agents less than 4 weeks before beginning the trial.
* Patients with asthma, angina pectoris or congestive heart failure.
* Patients with autoimmune disease such as lupus erythematosus, rheumatoid arthritis or thyroiditis.
* Patients with active infections including viral hepatitis.
* Patients with a history of any other neoplastic disease less than 5 years ago (carcinomas in situ of the cervix and basal/squamous cell carcinomas of the skin, however, can be admitted to the study).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-03; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the combination of DC vaccination and CPA therapy in human subjects | 2 Years
Feasibility of this combination therapy | 2 Years
Objective clinical responses | 2 Years

SECONDARY OUTCOMES:
Immunogenicity of DC vaccinations in subjects | 2 Years
Effect of CPA at this dose and schedule on the regulatory/suppressor T cells | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W. Fay, MD, Principal Investigator — Baylor Health Care System; Anna Karolina Palucka, MD, PhD, Study Director — Baylor Research Institute
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States